CLINICAL TRIAL: NCT01110135
Title: A Phase II Study of Bendamustine (B), Etoposide (E), Dexamethasone (D), and GCSF for Peripheral Blood Hematopoietic Stem Cell Mobilization (BED)
Brief Title: Bendamustine Hydrochloride, Etoposide, Dexamethasone, and Filgrastim For Peripheral Blood Stem Cell Mobilization in Treating Patients With Refractory or Recurrent Lymphoma or Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ajay Gopal, Principal Investigator, University of Washington
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 7176; NCI-2010-00509 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-04-20; First posted 2010-04-26 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-04

CONDITIONS: Adult Nasal Type Extranodal NK/T-cell Lymphoma; Anaplastic Large Cell Lymphoma; Angioimmunoblastic T-cell Lymphoma; Cutaneous B-cell Non-Hodgkin Lymphoma; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Intraocular Lymphoma; Nodal Marginal Zone B-cell Lymphoma; Peripheral T-cell Lymphoma; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Grade III Lymphomatoid Granulomatosis; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Adult T-cell Leukemia/Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Multiple Myeloma; Small Intestine Lymphoma; Splenic Marginal Zone Lymphoma; Waldenström Macroglobulinemia
MeSH Terms: conditions — Lymphoma, Extranodal NK-T-Cell; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Intraocular Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, T-Cell, Peripheral; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Multiple Myeloma; Waldenstrom Macroglobulinemia | interventions — Bendamustine Hydrochloride; Dexamethasone; Calcium Dobesilate; Filgrastim; Granulocyte Colony-Stimulating Factor; Leukapheresis; Flow Cytometry; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (chemotherapy and colony-stimulating factor) (Experimental): Patients receive bendamustine hydrochloride IV over 30-60 minutes on days 1 and 2, etoposide IV over 60-240 minutes on days 1-3, dexamethasone PO on days 1-4, and filgrastim SC beginning on day 5 and continuing until peripheral blood stem cell collection is complete. Patients undergo leukapheresis daily for a minimum of 3 days or until > 5 x 10^6 CD34+/kg has been collected.
  .
  Interventions: Drug: bendamustine hydrochloride; Drug: dexamethasone; Biological: filgrastim; Procedure: leukapheresis; Other: laboratory biomarker analysis; Other: flow cytometry; Drug: etoposide

INTERVENTIONS:
Drug: bendamustine hydrochloride — Given IV
  Other Names: bendamustin hydrochloride; bendamustine; cytostasan hydrochloride; Treanda
Drug: dexamethasone — Given PO
  Other Names: Aeroseb-Dex; Decaderm; Decadron; DM; DXM
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Procedure: leukapheresis — Given IV
Other: laboratory biomarker analysis — Correlative studies
Other: flow cytometry — Correlative studies
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213

SUMMARY:
This phase II trial is studying how well giving bendamustine hydrochloride, etoposide, dexamethasone, and filgrastim together for peripheral stem cell mobilization works in treating patients with refractory or recurrent lymphoma or multiple myeloma. Giving chemotherapy, such as bendamustine hydrochloride, etoposide, and dexamethasone, before a peripheral stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. Giving colony-stimulating factors, such as filgrastim, and certain chemotherapy drugs helps stem cells move from the bone marrow to the blood so they can be collected and stored

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the frequency of bendamustine (bendamustine hydrochloride) combined with GCSF (filgrastim) and dexamethasone to successfully mobilize peripheral blood stem cells (PBSCs) (as determined by collecting a minimum of 2 x 10^6 cluster of differentiation (CD)34+/kg).

SECONDARY OBJECTIVES:

I. To evaluate the response rate to bendamustine by diagnosis using established disease-specific response criteria.

II. To examine the number of apheresis cycles required to collect a minimum of 2 x 10^6 CD34+ cells/kg and ideally >= 5 x 10^6 CD34+ cells/kg (when achievable).

III. To assess the impact of bendamustine on B and T-lymphocyte populations in the peripheral blood (CD20+ cells, natural killer [NK] cells, CD4+25+ foxP3- regulatory cells, and CD8 cells).

OUTLINE:

Patients receive bendamustine hydrochloride intravenously (IV) over 30-60 minutes on days 1 and 2, etoposide IV over 60-240 minutes on days 1-3, dexamethasone orally (PO) on days 1-4, and filgrastim subcutaneously (SC) beginning on day 5 and continuing until peripheral blood stem cell collection is complete. Patients undergo leukapheresis daily for a minimum of 3 days or until > 5 x 10^6 CD34+/kg has been collected.

After completion of study treatment, patients are followed for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have relapsed or primary refractory lymphoid malignancy (including B-cell, T-cell, or Hodgkin lymphoma), or multiple myeloma; other transplant eligible diagnoses (e.g. germ cell tumor) can be included with principal investigator (PI) approval
* World Health Organization (WHO) classification of patients' malignancies must be provided
* Patients with lymphoid malignancies must have a computed tomography (CT) of chest, abdomen, and pelvis within six weeks of enrollment; patients with evidence of lymphadenopathy in the neck must have a CT of neck
* Patients must have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelets >= 100,000/mm^3 (without transfusion or growth factor support)
* Creatinine clearance (CrCl) greater than 50/ml per minute (all tests must be performed within 28 days prior to registration)
* Total bilirubin < 1.5 times upper limit of normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 times upper limit of normal
* All patients must be informed of the investigational nature of this study and have given written consent in accordance with institutional and federal guidelines
* Adequate venous access plan in place for apheresis procedure
* Three or fewer prior myelotoxic treatment regimens (specific regimens include ifosfamide, carboplatin and etoposide [ICE]; cisplatin, cytarabine, and dexamethasone [DHAP]; methotrexate [MTX]/high-dose cytarabine [HiDAC]; cyclophosphamide, vincristine, doxorubicin, and dexamethasone [hyperCVAD]; bortezomib, thalidomide, dexamethasone and 4-day continuous infusions of cisplatin, doxorubicin, cyclophosphamide, and etoposide [VTD-PACE])

Exclusion Criteria:

* Patients known positive for human immunodeficiency virus (HIV), or infectious hepatitis type B or C
* Pregnant or nursing women; men or women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Greater than six prior cycles of lenalidomide therapy
* Patients who have previously demonstrated resistance to bendamustine therapy (i.e. no response or progression w/in 6 months)
* Fludarabine or other nucleoside analog (except gemcitabine or cytarabine) therapy within 24 months of registration; patients with limited exposure to fludarabine/other nucleoside analog therapy within 24 months may be considered eligible with review and approval by the PI or Co-PI prior to study entry
* Symptomatic cardiopulmonary disease
* Prior autologous or allogeneic transplantation
* Prior radioimmunotherapy within 12 weeks of registration
* Prior failed (< 5 x 10^6 CD34/kg) PBSC collection due to inability to mobilize stem cells
* Prior pelvic or spinal irradiation
* Previous systemic chemotherapy/immunotherapy within 3 weeks before study entry
* Concurrent use of other anti-cancer agents or experimental treatments
* Known allergy or intolerance to bendamustine, mannitol, GCSF or dexamethasone
* More than 3 cycles of myelotoxic salvage chemotherapy within the past 4 months (specific regimens include ICE, DHAP, MTX/HiDAC, hyperCVAD, VTD-PACE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-08; Primary Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay Gopal, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Chemotherapy and Colony-stimulating Factor): Patients receive bendamustine hydrochloride IV over 30-60 minutes on days 1 and 2, etoposide IV over 60-240 minutes on days 1-3, dexamethasone PO on days 1-4, and filgrastim SC beginning on day 5 and continuing until peripheral blood stem cell collection is complete. Patients undergo leukapheresis daily for a minimum of 3 days or until > 5 x 10^6 CD34+/kg has been collected.
  .
  bendamustine hydrochloride: Given IV
  dexamethasone: Given PO
  filgrastim: Given SC
  leukapheresis: Given IV
  laboratory biomarker analysis: Correlative studies
  flow cytometry: Correlative studies
  etoposide: Given IV
Period: Overall Study
Arm/Group | Treatment (Chemotherapy and Colony-stimulating Factor)
Started | 43
Completed | 34
Not Completed | 9

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Chemotherapy and Colony-stimulating Factor)
Number analyzed (Participants) | 34
Age, Continuous [Median (Full Range); unit: years] | 61 [46 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Successful Mobilization and Collection of PBSCs
Description: Count of participants with successful mobilization and collection of PBSCs. Defined as collection of > 2 x 10^6 CD34/kg. The current study will be deemed to be potentially efficacious if the observed rate of success is at least 80%.
Time Frame: Within 7 days of apheresis and within 6 weeks of receiving bendamustine hydrochloride
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Chemotherapy and Colony-stimulating Factor)
Number analyzed (Participants) | 34
Participants | 34

ADVERSE EVENTS:
Arm/Group | Treatment (Chemotherapy and Colony-stimulating Factor)
Serious Adverse Events (participants affected / at risk) | 6/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Chemotherapy and Colony-stimulating Factor) (N=34)
Hypotension (Vascular disorders) | 2
Stroke (Nervous system disorders) | 1
Renal insufficiency (Renal and urinary disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Neutropenic fever (Blood and lymphatic system disorders) | 1
Sepsis (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Chemotherapy and Colony-stimulating Factor) (N=34)
Lymphopenia (Blood and lymphatic system disorders) | 34
Thrombocytopenia (Blood and lymphatic system disorders) | 31
Neutropenia (Blood and lymphatic system disorders) | 33
Leukopenia (Blood and lymphatic system disorders) | 26
Hypophosphatemia (Metabolism and nutrition disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 2
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Hypotension (Vascular disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes